CLINICAL TRIAL: NCT01695954
Title: The Effect of Efavirenz and Ritonavir-boosted Darunavir on the Pharmacokinetics of the HMG CoA Reductase Inhibitor Pitavastatin
Brief Title: Pharmacokinetic Study of Pitavastatin and Ritonavir-Boosted Darunavir or Efavirenz
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York City Health and Hospitals Corporation (Other); Kowa Pharmaceuticals America, Inc. (Industry); University at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11-01787
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Hyperlipidemia; HIV
Keywords: HIV; Hyperlipidemia; Pharmacokinetics; Statins; Darunavir; Efavirenz; Pitavastatin
MeSH Terms: conditions — Hyperlipidemias | interventions — pitavastatin; Darunavir; Ritonavir; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Subjects assigned to Arm A will receive pitavastatin 2 mg at bedtime and efavirenz 600 mg at bedtime.
  Interventions: Drug: Pitavastatin; Drug: Efavirenz
- Arm B (Experimental): Subjects assigned to Arm B will receive pitavastatin 2 mg daily and darunavir 800 mg with ritonavir 100 mg daily.
  Interventions: Drug: Pitavastatin; Drug: Darunavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin 2 mg tablets taken at bedtime in Arm A and in the morning in Arm B.
  Other Names: Livalo
Drug: Darunavir — Darunavir 400 mg tablets x 2 taken daily in Arm B
  Other Names: Prezista
  Arms: Arm B
Drug: Ritonavir — Ritonavir 100 mg tablets taken daily in Arm B
  Other Names: Norvir
  Arms: Arm B
Drug: Efavirenz — Efavirenz 600 mg tablets taken at bedtime in Arm A
  Other Names: Sustiva
  Arms: Arm A

SUMMARY:
The main goal of this study is to determine how taking efavirenz affects the levels of pitavastatin in the bloodstream when both drugs are taken together and to see how darunavir with ritonavir affects the levels of pitavastatin in the bloodstream. Secondary goals are to see how taking pitavastatin affects the levels in the blood of efavirenz when both drugs are taken together and to see how taking pitavastatin affects the levels in the blood of darunavir.

DETAILED DESCRIPTION:
HIV infected persons are at risk for coronary heart disease due to chronic inflammation associated with the virus itself, the side effects of the antiretroviral (ARV) therapies which can cause elevated cholesterol, and the risk factors such as smoking, high blood pressure and family history of heart disease.

The most commonly prescribed ARVs for treatment of HIV are efavirenz and drugs in the protease inhibitor (PI) class such as darunavir with ritonavir. To treat elevated cholesterol in patients infected with HIV, guidelines recommend the use of statins (a class of lipid lowering drugs). PIs and efavirenz can increase the levels of some statins and reduce the levels of others in the bloodstream. Pitavastatin (Livalo) is a statin approved by the Food and Drug Administration (FDA) for the treatment of high cholesterol.

In order to be able to use pitavastatin safely in HIV-infected patients taking either darunavir with ritonavir or efavirenz, it is important to study how taking pitavastatin with darunavir and ritonavir or pitavastatin with efavirenz affect the levels of each of these drugs in the bloodstream.

Twenty-eight participants will be enrolled in one of two study arms: 14 in Arm A and 14 in Arm B.

Arm A:

Participants will start taking pitavastatin 2 mg tablets every night at bedtime. On day 4 participants will come in for a 14-hour pharmacokinetic (PK) overnight visit and will have about 9 tablespoons of blood drawn. Participants will return 12 hours after the last blood draw for a final blood draw. They will then stop taking pitavastatin. Participants will then start taking one efavirenz 600 mg tablet at bedtime.

On day 14, participants will come in for a second 14-hour visit and will have about 9 tablespoons of blood drawn. They will return 12 hour after the last blood draw for a final blood draw. Participants will then start taking both pitavastatin and efavirenz at bedtime.

On day 18, participants will come in for a third 14-hour PK visit and will have about 9 tablespoons of blood drawn. They will return 12 hour after the last blood draw for a final blood draw. They will then stop taking all study drugs and will either come in or receive a final phone call on day 25.

Arm B:

Participants will start taking one pitavastatin 2 mg tablet every morning. On day 4 participants will come in for a 14-hour pharmacokinetic (PK) daytime visit and will have about 9 tablespoons of blood drawn. Participants will return 12 hours after the last blood draw for a final blood draw. They will then stop taking pitavastatin. Participants will then start taking darunavir 400 mg tablets (2) and ritonavir 100 mg tablets (1) every morning.

On day 14, participants will come in for a second 14-hour visit and will have about 9 tablespoons of blood drawn. They will return 12 hour after the last blood draw for a final blood draw. Participants will then start taking one pitavastatin 2mg tablet, two darunavir 400 mg tablets and one ritonavir 100 mg tablet.

On day 18, participants will come in for a third 14-hour PK visit and will have about 9 tablespoons of blood drawn. They will return 12 hour after the last blood draw for a final blood draw. They will then stop taking all study drugs and will either come in or receive a final phone call on day 25.

ELIGIBILITY:
Inclusion Criteria:

* Absence of HIV-1 infection as documented by any licensed ELISA test kit within 21 days prior to study entry.
* Male or female aged 18-60 years.
* Able and willing to provide informed consent.
* All men and women of reproductive potential must practice adequate birth control to prevent pregnancy from start of the study until completion of the study.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to study entry and day of entry.
* Hemoglobin > 12.5 g/dL for men; > 11.5 g/dL for women;
* Absolute neutrophil count >1,500 cells/mm3;
* Platelet count > 100,000 platelets/mm3;
* AST (SGOT)/ALT (SGPT) <1.5X ULN;
* Creatinine <1.5 X ULN
* Subject is within 20% (+/-) of ideal body weight and must weigh at least 50 kg

Exclusion Criteria:

* Use of illicit drugs or alcohol which would interfere with the completion of this study.
* Pregnancy or breast-feeding.
* History of chronic illnesses such as hypertension, coronary artery disease, arthritis, diabetes, or any chronic gastrointestinal conditions which might interfere with drug absorption.
* Any medical condition which, in the opinion of the investigator, would interfere with the subjects ability to participate in this protocol.
* Use of prohibited protocol-specified drugs, prescription or over-the-counter within 14 days prior to study entry.
* Participation in any investigational drug studies within 30 days prior to study entry.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Aberg, M.D., Principal Investigator — NYU School of Medicine
Locations (1):
- Bellevue/NYU AIDS Clinical Trials Unit, New York, New York, United States

REFERENCES:
- [Result] Malvestutto CD, Ma Q, Morse GD, Underberg JA, Aberg JA. Lack of pharmacokinetic interactions between pitavastatin and efavirenz or darunavir/ritonavir. J Acquir Immune Defic Syndr. 2014 Dec 1;67(4):390-6. doi: 10.1097/QAI.0000000000000333. PMID 25202920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual began August 24, 2012 and ended January, 8, 2013. All study procedures took place at the NYU/Bellevue Clinical Trials Unit and NYU Clinical and Translational Science Institute.
Groups:
- Arm A: (Pitavastatin and Efavirenz): Subjects assigned to Arm A will receive pitavastatin 2 mg at bedtime and efavirenz 600 mg at bedtime.
- Arm B: (Pitavastatin and Ritonavir-boosted Darunavir): Subjects assigned to Arm B will receive pitavastatin 2 mg daily and darunavir 800 mg with ritonavir 100 mg daily.
Period: Overall Study
Arm/Group | Arm A: (Pitavastatin and Efavirenz) | Arm B: (Pitavastatin and Ritonavir-boosted Darunavir)
Started | 18 | 16
Completed | 14 | 14
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: (Pitavastatin and Efavirenz) | Arm B: (Pitavastatin and Ritonavir-boosted Darunavir) | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 16 | 34
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: 24-hour area under the curve (AUC) for pitavastatin when coadministered with efavirenz and with darunavir/ritonavir and 24-hour AUC for efavirenz or darunavir when coadministered with pitavastatin
Time Frame: 0 to 24 hours
Population: Subjects who completed all visits
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Arm A: (Pitavastatin and Efavirenz): Subjects assigned to Arm A will receive pitavastatin 2 mg at bedtime for the first 4 days, then efavirenz 600 mg at bedtime for the next 10 days and both pitavastatin 2 mg and efavirenz 600 mg at bedtime for the final 4 days. Blood will be drawn on days 0, 4, 14 and 18.
- Arm B: (Pitavastatin and Darunavir): Subjects in arm will receive pitavastatin 2 mg daily for the first 4 days, then darunavir 400 mg x 2 tabs and ritonavir 100 mg x 1 tab daily for the next 10 days and will receive both pitavastatin 2 mg and darunavir 400 mg x 2 tabs and ritonavir 100 mg x 1 tab daily for the final 4 days. Blood will be drawn on days 0, 4, 14, and 18.
Arm/Group | Arm A: (Pitavastatin and Efavirenz) | Arm B: (Pitavastatin and Darunavir)
Number analyzed (Participants) | 18 | 16
ng*hr/mL | 85.3 (5.72) | 62.8 (6.24)

2. Secondary Outcome: GMR of Cmax of Pitavastatin When Coadministered With Efavirenz or With Darunavir/Ritonavir
Description: Geometric Mean Ratio (GMR) of Cmax for pitavastatin with Efavirenz vs. alone and GMR of Cmax for pitavastatin with darunavir/ritonavir vs. alone was reported.
Time Frame: Day 18
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Arm A: (Pitavastatin and Efavirenz) | Arm B: (Pitavastatin and Ritonavir-boosted Darunavir)
Number analyzed (Participants) | 18 | 16
ng/mL | 1.20 [0.79 to 1.83] | 0.93 [0.72 to 1.19]

3. Primary Outcome: GMR of 24- Hour AUC of Pitavastatin When Coadministered With Efavirenz or With Darunavir/Ritonavir Over 24 Hour AUC of Pitavastatin
Description: Geometric Mean Ratio (GMR) of 24- Hour Area under the plasma drug concentration-time curve (AUC) of pitavastatin when coadministered with efavirenz or with darunavir/ritonavir over 24 Hour (AUC) of pitavastatin
Time Frame: 0 to 24 hours
Population: Subjects who completed all visits
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Arm A: (Pitavastatin and Efavirenz) | Arm B: (Pitavastatin and Darunavir)
Number analyzed (Participants) | 18 | 16
Ratio
  GMR of Pitavastatin with (EFV or DRV)/Pitavastatin | .89 [.7321 to 1.09] | .91 [.78 to 1.06]
  GMR of (EFV or DRV) with Pitavastatin/(EFV or DRV) | .90 [.75 to 1.06] | 1.08 [.96 to 1.22]

ADVERSE EVENTS:
Time Frame: 7 months.
Arm/Group | Arm A: (Pitavastatin and Efavirenz) | Arm B: (Pitavastatin and Ritonavir-boosted Darunavir)
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 14/18 | 7/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: (Pitavastatin and Efavirenz) (N=18) | Arm B: (Pitavastatin and Ritonavir-boosted Darunavir) (N=16)
Headache (Nervous system disorders) | 2 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0)
Nausea (Nervous system disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vivid dreams (Nervous system disorders) | 1 (2) | 0 (0)
Pain at venipuncture site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CPK elevation (General disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Pitavastatin levels for 4 subjects enrolled in Arm B were lost due to emergency transfer of specimens to temporary storage facility during Hurricane Sandy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No